CLINICAL TRIAL: NCT01176214
Title: Weaning by Early Versus lAte Tracheostomy iN supratentorIal iNtracerebral Bleedings
Brief Title: WEANING-Study: "Weaning by Early Versus lAte Tracheostomy iN supratentorIal iNtracerebral Bleedings
Acronym: WEANING
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment of patients
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WEANING-Study2010
Record Dates: First submitted 2010-07-26; First posted 2010-08-05 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Intracerebral Hemorrhage
Keywords: supratentorial intracerebral hemorrhage; tracheostomy; sedation; weaning
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- early tracheostomy (Experimental): see study description
  Interventions: Procedure: Early tracheostomy
- late tracheostomy (Active Comparator): Compared to the "early tracheostomy"-group, those patients who have been randomized to "late tracheostomy" will undergo conventional tracheostomy between day 12 - 14 if extubation fails
  Interventions: Procedure: Late tracheostomy

INTERVENTIONS:
Procedure: Early tracheostomy — Patients with supratentorial ICH who require mechanical ventilation, fulfill the inclusion criteria, and have been randomized to the "treatment arm" will receive an early tracheostomy within 72h after symptom onset.
  Arms: early tracheostomy
Procedure: Late tracheostomy — Compared to the "early tracheostomy"-group, those patients who have been randomized to "late tracheostomy" will undergo conventional tracheostomy between day 12 - 14 if extubation fails
  Arms: late tracheostomy

SUMMARY:
Background:

One third of all ICH patients require intubation and mechanical ventilation and 1/3 of all ventilated patients require tracheostomy (i.e.≈10% of all ICH patients require tracheostomy). As shown previously, predisposing factors for tracheostomy are hematoma volume, hemorrhage location, presence of intraventricular hemorrhage (IVH), and occlusive hydrocephalus as well as presence of COPD (Huttner HB et al 2006 CVD).

Sustained restricted vigilance and impaired consciousness after ICH is likely to result in failure of extubation, raise in incidence of ventilator-associated pneumonia, increased amount of sedative drugs and prolonged duration of neurocritical care.

Hence an early tracheostomy may be beneficial in terms of reduced duration of mechanical ventilation.

Basic hypothesis:

Compared to patients with conventional ("late") tracheostomy between day 12 - 14, patients with "early" tracheostomy within 72h after admission will have:

* shorter cumulative time of mechanical ventilation
* less incidence of ventilator-associated pneumonia
* less consumption of sedative drugs
* shorter duration of stay in neurocritical care unit

Randomization:

Consecutive eligible patients are randomly assigned to Either "early" tracheostomy within 72h after hospital admission Or "late" tracheostomy (= control group; undergoing conventional tracheostomy between day 12 - 14 if extubation fails) Both groups receive plastic tracheostomy

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring intubation / mechanical ventilation
* Supratentorial intracerebral hemorrhage (including:)
* primary spontaneous ICH (lobar / deep)
* ICH related to anticoagulant therapy
* with or without intraventricular hemorrhage
* with or without occlusive and / or communicating hydrocephalus
* Hematoma volume >0 ml and <60 ml
* Age 18 - 85 years
* Informed consent (legal representative)

Exclusion Criteria:

* Patients with elective intubation/ventilation for EVD placement
* Patients with "do not treat" / "do not resuscitate" orders, severe co- morbidity and life expectancy of less than 3 months
* Absent consent of relatives for invasive (neuro-)critical care
* Contraindication for tracheostomy
* Other than primary supratentorial ICH or supratentorial ICH related to oral anticoagulants
* Pre-existing COPD (known/treated)
* Pre-existing congestive heart failure (≥3 NYHA)
* Pre-existing modified Rankin Scale (≥4)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cumulative time requiring mechanical ventilation and Overall duration of neurocritical care | 30 days
  Primary End-points:
  * Cumulative time requiring mechanical ventilation
  * Overall duration of neurocritical care

SECONDARY OUTCOMES:
Incidence of respirator-associated pneumonia | 30 days
Cumulative consumption of sedative drugs | 30 days
Incidence of episodes with increased intracranial pressure | 30 days
In-hospital mortality | 30 days
3-months functional outcome (mRS) | 90 days
  functional outcome after 3 months using the modified Rankin Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hagen B Huttner, MD, Principal Investigator — Department of Neurology, University of Erlangen-Nuremberg, Germany; Martin Köhrmann, MD, Study Director — Department of Neurology, University of Erlangen, Germany; Dimitre Staykov, MD, Study Director — Department of Neurology, University of Erlangen, Germany
Locations (1):
- University or Erlangen-Nuremberg, Erlangen, Germany